CLINICAL TRIAL: NCT04804462
Title: Virtual Reality Meditation for Fatigue in Persons With Rheumatoid Arthritis
Brief Title: Virtual Reality Meditation for Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Nathan Dreesmann, Registered Nurse, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00007661; TL1TR002318 (NIH)
Record Dates: First submitted 2019-07-02; First posted 2021-03-18 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Fatigue; Rheumatoid Arthritis
Keywords: mindfulness; distraction; chronic pain; mixed methods; outpatient
MeSH Terms: conditions — Fatigue; Arthritis, Rheumatoid; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This study will employ a convergent mixed-methods design with quantitative and qualitative data collection occurring concurrently throughout the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Meditation for Fatigue (Experimental): Participants will experience Virtual Reality Meditation in the comfort of their own home.
  Interventions: Device: Virtual Reality Meditation

INTERVENTIONS:
Device: Virtual Reality Meditation — After donning the VR headset, participants will be able to use a handheld controller to choose from several virtual outdoor settings, three types of meditation, and three session lengths. After choosing their desired option, participants will experience virtual reality meditation in the desired virtual location, of the desired meditation type, and for the allotted duration chosen.

SUMMARY:
This study will examine the feasibility and acceptability of using virtual reality (VR) meditation to manage fatigue in outpatients with rheumatoid arthritis (RA). The specific aims of this feasibility study include: 1) examining the feasibility of implementing VR meditation as an adjunct for managing fatigue in outpatients with rheumatoid arthritis; 2) determine the acceptability of using VR-delivered meditation training for fatigue management in outpatients with rheumatoid arthritis; and 3) is to explore outpatient's experience of using VR-delivered meditation to manage fatigue.

DETAILED DESCRIPTION:
RA is a debilitating disease that affects over 1.3 million people in the U.S. While recent advances in medicine have enhanced management of the disease, a staggeringly large portion of outpatients with RA still suffer from fatigue. A profound, unrelenting exhaustion affecting energy, motivation, and concentration, fatigue often develops over time without an inciting event. Fatigue includes complex interactions between physiological, psychological, and behavioral processes, making it not only insidious, but difficult to treat. Being multifaceted, fatigue impacts depression, mood, and physical activity, and can be exacerbated by pain, and current treatment options target each of these correlates of fatigue. Meditation has been extensively and effectively utilized in RA and other rheumatic diseases, yet, to date, VR meditation has yet to be deployed in this population.

This feasibility study will employ a mixed-methods design. Thirty adult outpatients with clinically-diagnosed rheumatoid arthritis will be enrolled from a local rheumatology clinic and utilize VR in their own home. Donning an Oculus Quest VR headset and using two handheld controllers, patients will have the opportunity to choose from several virtual outdoor settings, three types of meditation, and three session lengths. PROMIS measures of fatigue, depression, mood, pain, and physical activity will be collected at baseline and weekly intervals for the first 4 weeks, after which, an eight-week follow-up measure will be taken. Semi-structured patient interviews will be used to capture patient's experience of RA, fatigue, as well as experience of the virtual environment. This feasibility study's results will address the acceptability, desirability, implementation, practicality, adaptation, integration, expansion, and "limited" efficacy testing of utilizing VR meditation for managing fatigue in outpatients with RA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of rheumatoid arthritis

Exclusion Criteria:

* Individuals with a past medical history of uncorrectable visual or auditory impairment, history of seizure disorder or seizure caused by technology use, extensive motion sickness, vestibular dysfunction, severe neck immobility, or excessive face or scalp sensitivity to pressure. These criteria were chosen as immersion and presence necessitate sufficient vision and hearing, technology use may cause side effects in persons with seizure history, severe motion sickness or vestibular dysfunction, neck immobility may decrease immersion and presence, and scalp sensitivity may inhibit use of a head-mounted device (HMD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of Using Virtual Reality Meditation | 4 weeks
  Completion percentage of quantitative questionnaires and an analysis of fidelity will provide insight into the feasibility of using virtual reality meditation for rheumatoid-arthritis related fatigue.
Acceptability of Using Virtual Reality Meditation | 4 weeks
  Qualitative interviews, paired with quantitative questionnaires, will inform the acceptability of both study procedures and measures of fatigue, anxiety, depression, pain behavior, physical functioning, and mood for use in outpatients with rheumatoid-arthritis.
Experience of Using Virtual Reality Meditation | 4 weeks
  Qualitative interviews will aid exploration of participant's experience of using virtual reality meditation for rheumatoid-arthritis related fatigue.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.0 - Fatigue | 4 weeks
  Scores Range: 0-100; Uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  On the T-score metric, a score of 40 is one SD lower than the mean of the reference population and a score of 60 is one SD higher than the mean of the reference population.
  PROMIS measures are scored on the T-score metric. High scores mean more of the concept being measured. PROMIS measures for fatigue will be deployed using a computer-adaptive test (CAT) that will be emailed to participants. More information from: https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis
Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.0 - Depression | 4 weeks
  Scores Range: 0-100; Uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  On the T-score metric, a score of 40 is one SD lower than the mean of the reference population and a score of 60 is one SD higher than the mean of the reference population.
  PROMIS measures are scored on the T-score metric. High scores mean more of the concept being measured. PROMIS measures for fatigue will be deployed using a computer-adaptive test (CAT) that will be emailed to participants. More information from: https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis
Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.0 - Anxiety | 4 weeks
  Scores Range: 0-100; Uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  On the T-score metric, a score of 40 is one SD lower than the mean of the reference population and a score of 60 is one SD higher than the mean of the reference population.
  PROMIS measures are scored on the T-score metric. High scores mean more of the concept being measured. PROMIS measures for fatigue will be deployed using a computer-adaptive test (CAT) that will be emailed to participants. More information from: https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis
Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.0 - Pain Behavior | 4 weeks
  Scores Range: 0-100; Uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  On the T-score metric, a score of 40 is one SD lower than the mean of the reference population and a score of 60 is one SD higher than the mean of the reference population.
  PROMIS measures are scored on the T-score metric. High scores mean more of the concept being measured. PROMIS measures for fatigue will be deployed using a computer-adaptive test (CAT) that will be emailed to participants. More information from: https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis
Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.2 - Physical Function | 4 weeks
  Scores Range: 0-100; Uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  On the T-score metric, a score of 40 is one SD lower than the mean of the reference population and a score of 60 is one SD higher than the mean of the reference population.
  PROMIS measures are scored on the T-score metric. High scores mean more of the concept being measured. PROMIS measures for fatigue will be deployed using a computer-adaptive test (CAT) that will be emailed to participants. More information from: https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis
Brief Mood Introspection Scale (BMIS) Scored | 4 weeks
  The BMIS will be deployed using a computer-adaptive test (CAT) that will be emailed to participants.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan J Dreesman, PhD, RN, Principal Investigator — University of Washington
Locations (1):
- Rheumatology Clinic at UW Medical Center - Roosevelt, Seattle, Washington, United States

REFERENCES:
- [Derived] Dreesmann NJ, Buchanan D, Tang HJ, Furness Iii T, Thompson H. Virtual Reality Meditation for Fatigue in Persons With Rheumatoid Arthritis: Mixed Methods Pilot Study. JMIR Form Res. 2023 Oct 17;7:e46209. doi: 10.2196/46209. PMID 37847542